CLINICAL TRIAL: NCT01213797
Title: Impact of the Suicide Attempt on the Close Entourage: Traumatic Stress and Medico-economic Concerns, in Medium and Long Term
Brief Title: IMTAP : Impact of the Suicide Attempt on the Nearly Entourage in Term of Traumatic Stress and Medico-economic Impact
Acronym: IMTAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: DGS 2006/0116; PHRC 2005/1917 (Other: DHOS); 2006/0603 (Other: Sponsor)
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-07

CONDITIONS: Suicide, Attempted; Relatives
Keywords: Suicide
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suicide attempter and its entourage: Suicide attempter and its close relatives (who are living under the same roof)
  Comparison of the population of the close relations of committing suicide with the data of the Research Institute and Documentation in Economy of Health (IRDES) on the French population (sample of 20.000 people, representative of 95% of the French households).

SUMMARY:
With 11.000 deaths and 150.000 attempts each year in France, the suicide represents an important public health problem. For each death by suicide, one can count 6 "direct" bereaved people and 20 people in more indirect connection with this mourning (Terra 2001). In term of impact, there is thus 300.000 people (annually) touched by the deaths by suicide and 3.750.000 people (annually) touched by the "suicide attempt" of a close relative. It seems indeed important to have Public Health data on this cascade repercussion of the suicide attempt.

A suicide attempt propagates a suffering cascade on the various circles of the family and close entourage, which can be measured in term of traumatic stress and medico-economic impact.

Objective = To measure the medico-economic impact on the entourage, in the 3 months following the suicide attempt and at 1 year.

DETAILED DESCRIPTION:
Secondary objectives = To measure the impact of the suicide attempt in traumatic term of stress on the close relatives of committing suicide confronted with the suicidal scene To compare the evolution of consumption of care of the close relatives and of committing suicide To measure the evolution of the general health condition of the close relatives and of committing suicide

The study participants (committing suicide it and the relatives) will be recontacted by telephone, after 3 months and to 1 year.

Consumption of care (number of consultations, drugs consumption) of the population of the close relatives of committing suicide will be compared with the data of the Research Institute and Documentation in Economy of Health (IRDES) on the French population (sample of 20.000 people, representative of 95% of the French households).

ELIGIBILITY:
Inclusion Criteria for Suicide attempter :

* Men or women
* Older than 18 years
* Survivor with an suicide attempt going back to less than 15 days

Inclusion Criteria for close relations of committing suicide :

* Men or women
* age more than 18 years
* Members of the entourage of committing suicide
* Living under the same roof as committing suicide it

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 500 families; 500 committing suicide and approximately 900 close relatives.
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2006-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Consumption of care in the close relatives of a suicide attempter | one year
  Consumption of care in the close relatives of a suicide attempter, at the various stages of evaluation, compared with a matched sample in general population (data IRDES). One will be able to thus evaluate not only if the consumption of the close relatives is higher than the average, but still if this difference increases or on the contrary decreases during time.

SECONDARY OUTCOMES:
Psychological level of distress | one year
  Psychological level of distress in the close relatives
Links between consumption of care and psychological level of distress | one year
  Links between consumption of care and psychological level of distress
Prevalence of the post-traumatic stress disorder | one year
  Post-traumatic stress disorder at 3 months and one year, as evaluated by the PTSD Check List Symptoms among members of the entourage having been exposed to the scene of the suicide attempt.
  Comparison of prevalence of the post-traumatic disorder of stress compared to the index of lethality of the suicide attempt index.
Evolution of consumption of care | one year
  Evolution of consumption of care at committing suicide compared to the remainder of the household and the general population

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume VAIVA, Principal Investigator — University Hospital, Lille
Locations (12):
- France (12):
  - University Hospital, Angers, Angers
  - University Hospital, Brest, Brest
  - University Hospital, Caen, Caen
  - University Hospital, Clermont-Ferrand, Clermont-Ferrand
  - University Hospital, Lille, Lille
  - University Hospital, Limoges, Limoges
  - Le Vinatier Hospital, Lyon
  - University Hospital, Nancy, Nancy
  - University Hospital, Nice, Nice
  - Tenon Hospital, Paris, Paris
  - General Hospital, Quimper, Quimper
  - EPSM Lille Metropole, Tourcoing